CLINICAL TRIAL: NCT05202392
Title: Effect of Myofascial Release With Isometric Exercise Versus Myofascial Release With Scapular Stabilization Exercise on Neck Pain in Young Adults With Text Neck Syndrome
Brief Title: Effects of Myofascial Release With Isometric Exercises Versus Scapular Stabilization Exercise on Neck Pain in Text Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-FSD-00242
Record Dates: First submitted 2022-01-08; First posted 2022-01-21 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Neck Pain
Keywords: text neck syndrome; pain and disability; isometrics; scapular stabilization; myofascial release
MeSH Terms: conditions — Neck Pain; Pain | interventions — Myofascial Release Therapy; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study will be single-blinded with blinding of the assessor to the groups and the therapist (researcher). After the initial screening process is completed, an independent accessor will access each recruited patient, outcome measuring tolls will be used by the experts. This will be recorded as baseline measurement assessment. The treatment will base on the designed protocol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial release with Isometric Exercises (Experimental): Myofascial release technique combined with isometric exercises will be given to first group. Patients in this group will be given muscle stretching along with trigger point release for following muscles. For the trapezius muscle as the patient will be in sitting and restrained friction for 30 seconds will be applied to a primary trigger point along with passive trapezius stretching on the alternative side. A chin tuck will be applied to stretch the sub-occipital muscles. Flexion and slight rotation of head will stretch the posterior rotator muscles. The extension of neck and its rotation will stretch sternocleidomastoid muscle. Combining lateral bend to alternative medial head will stretch the scalene muscles. Isometrics for this group will be neck flexion, isometric neck extension, isometric neck side flexion, Isometric neck rotation, neck extensors stretch, neck flexors and side flexors stretch, stretch for right side and lateral rotation stretch
  Interventions: Other: Myofascial release with isometric exercises
- Myofascial Release with Scapular Stabilization Exercise (Experimental): These individuals will only receive same myofascial release therapy as 1st group combined with stabilization exercises. The stabilization exercises will include total 5 stages. The patient will be instructed to get into a supine position and to relax their body and will be instructed to place their feet flat on floor while bending their knees and holding this posture without and involvement of neck movements. After this, the subjects will be taught to raise their shoulder arm up to 90° combined with full scapular protraction and elbow extension and to hold this position for 10 seconds before returning to the prior positions doing this for 3 laps and 10 repetitions and with a minute break in between. For a quadruped position the individuals will alternatively lift their arms along with 120° flexion and shoulder abduction and hold this for ten seconds for ten repetitions for 3 laps and a 30 second break in between
  Interventions: Other: Myofascial release with scapular stabilization exercise

INTERVENTIONS:
Other: Myofascial release with isometric exercises — Patients in group A will receive 40 minutes of combined therapy treatment session including myofascial release of muscles with trigger point release and 5 isometric exercises of neck at alternative 3 days/week for 4 weeks.
  Arms: Myofascial release with Isometric Exercises
Other: Myofascial release with scapular stabilization exercise — Patients in group B will get 40 minutes of myofascial therapy same as the first group combined with scapular stabilization exercise in 5 different positions and this treatment session will be at alternative 3 days/week for 4 weeks.
  Arms: Myofascial Release with Scapular Stabilization Exercise

SUMMARY:
The objective of this study is to investigate the effects of myofascial release combined with isometrics and with scapular stabilization on neck pain, disability and ROM in young adults with text neck syndrome

DETAILED DESCRIPTION:
Neck pain NP (pain in cervical region) has been a major issue these days related to the increased use of smartphones. A posture that has been developed by growing use of technology is a posture called the Text Neck, which has become an epidemic to the world. The text neck is a posture in which a person keeps their head down (forward head posture) to look at their device for long periods of time. There are many medications and techniques used in management of neck pain. Myofascial release has been proved to be efficacious for pain in the neck. This study is unique in that it examines the effect of myofascial therapy along with isometric exercises or scapular stabilization exercises on neck pain, disability, movements and daily life activities.

ELIGIBILITY:
Inclusion Criteria:

* Young adults including both female and male between the ages of 18 to 26 years with neck pain who were using smart phone, tablet or laptop for past six-month duration and above.
* Subjects with average 3 or more than 3 hours mobile usage and who may have 3 out of the 6 possible symptoms for text neck which include pain in neck, upper back and shoulder pain, headache as well as insomnia, tingling and numbness in the hands for more than 6 months and with a complain of pain in neck after use of mobile phones or other gadgets.
* Individuals with NDI score of minimum 30%-48% i.e., moderate disability.
* Individuals with willingness to participate in this study.

Exclusion Criteria:

* Specific causes of neck pain involving problems including neurological involvement such as myelopathy combined with weakness, sensory loss with numbness, cervical spinal stenosis and prolapse.
* Any previous neck or upper limb surgery.
* Any neurological disorders including headache and irradiated pain due to some diagnosed disease with involvement of infection and malignancy
* Cerebrovascular insufficiency, carcinoma or traumatic fractures or any chronic disease of musculoskeletal system such as polyarthritis.
* Individuals with acute pain and inflammation, torticollis, acute osteoarthritis, vertigo, heart disease, pregnancy will be excluded from this research.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 2 months
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms such as pain
Neck Disability Index | 2 months
  The Neck Disability Index (NDI) is designed to measure neck-specific disability. The questionnaire has 10 items concerning pain and activities of daily living including personal care, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No